CLINICAL TRIAL: NCT04165902
Title: Additional Therapeutic Effects of Triamcinolone to Hyaluronic Acid on Knee Osteoarthritis: a Double-blind, Randomized-controlled Clinical Trial
Brief Title: Additional Effects of Steroid and Dextrose to Hyaluronic Acid on Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Professor, MD, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOST 108-2314-B-341-003
Record Dates: First submitted 2019-11-10; First posted 2019-11-18 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis, hyaluronic acid, steroid, dextrose
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- steroid plus hyaluronic acid (Experimental): steroid plus hyaluronic acid injection, one time per week, for 3 weeks
  Interventions: Drug: compare the effects of steroid plus hyaluronic acid and destrose plus hyaluronic acid on knee osteroarthritis
- dextrose plus hyaluronic acid (Active Comparator): dextrose plus hyaluronic acid injection, one time per week, for 3 weeks
  Interventions: Drug: compare the effects of steroid plus hyaluronic acid and destrose plus hyaluronic acid on knee osteroarthritis

INTERVENTIONS:
Drug: compare the effects of steroid plus hyaluronic acid and destrose plus hyaluronic acid on knee osteroarthritis — compare the immediate effect (one week after 3 times of injections), short-term effects (one month and three months after 3 times of injections), and midterm effect (6 months after 3 times of injections).

SUMMARY:
Using double-blind, randomized controlled design to compare the immediate, short-term and intermediate-term additional therapeutic effects of ultrasound-guided corticosteroid injection and dextrose injection of hyaluronic acid injection on patients with knee osteoarthritis, under the basis of International Classification of Functioning, Disability, and Health.

DETAILED DESCRIPTION:
A total of 60 patients will be collected. The participants will be randomized into two groups, including hyaluronic acid combined corticosteroid group and hyaluronic acid combined dextrose group. The balance, physical activity (10 meters normal and fast walk, up and downstairs, and 5 repeated chair-rising time, timed up and go test), functional performance and knee-related quality of life (Western Ontario and McMaster Universities Osteoarthritis index、Knee Injury and Osteoarthritis Outcome Score) will be evaluated. All the evaluations will be re-evaluated at one week after injection, one month after injection, three months after injection, and six months after injection. Subjects and evaluators will be both blinded to the group's classification during the whole course of study.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of knee osteoarthritis can walk for 15 meters Kellgren-Lawerence grade 2 or greater than 2 can follow up for 6 months

Exclusion Criteria:

* major diseases will affect balance, such as stroke, infectious diseases, rheumatoid arthritis, dizziness, or vertigo fractures malignance pregnancy or prepare to pregnant received knee injections in the past 6 months previous operation of knee joints

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-11 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis index | changes of scores from baseline to at one week, one month, 3 months and 6 months after 3 times of injections; score range: 0-100, higher scores mean a worse outcome
  assess knee osteoarthritis related performance

SECONDARY OUTCOMES:
Balance | changes of scores from baseling to at one week, one month, 3 months and 6 months after 3 times of injections; score range 0-4, higher scores mean a better outcome
  Berg Balance scale
physical functional performance-walking | change from baseline to at one week, one month, 3 months and 6 months after 3 times of injections
  10 meters normal and fast walking speed
physical functional performance-stairs climbing | change from baseline to at one week, one month, 3 months and 6 months after 3 times of injections
  time for up and down stairs
physical functional performance-chair raising | change from baseline to at one week, one month, 3 months and 6 months after 3 times of injections
  5 repeated chair-rising time
physical functional performance-balance | change from baseline to at one week, one month, 3 months and 6 months after 3 times of injections
  timed up and go test
Knee Injury and Osteoarthritis Outcome Score | changes of scores from baseline to at one week, one month, 3 months and 6 months after 3 times of injections; score range 0-100, higher scores mean at better outcome
  assess osteoarthritis of knee related function
Doppler resistance index | changes of scores from baseline to at one week after 1 time of injection and two weeks after 2 times of injection; the lower values indicate a low blood vessel resistance
  assess knee blood vessel resistance

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Study Chair — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No